CLINICAL TRIAL: NCT04424329
Title: Effect of a Specific Blend of Fibers and Probiotics on the Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19.17.NRC
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Microbiota Perturbation by an Environmental Challenge
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition intervention (Experimental): Ingestion of fibers and probiotics daily for 22 days
  Interventions: Dietary Supplement: Fibers and probiotics
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Fibers and probiotics — A blend of fibers and seven probiotics
  Arms: Nutrition intervention

SUMMARY:
The study will investigate the effect of a mix of fibers and probiotics on faecal microbiota challenged by an environmental stress

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed
2. Adult men and women aged 18 to 45 years
3. Healthy based on the medical screening visit and medical questionnaire
4. BMI in the range of 18.5 to 29.9 kg/m2.

Exclusion Criteria:

1. Known food allergy and intolerance
2. Currently participating in another clinical trial or research project
3. Fewer than 5 spontaneous bowel movements per week on average
4. Chronic or recurrent diarrhea with spontaneous bowel movements more often than 2 times daily
5. Systemic antibacterial/antifungal therapy during the 3 months prior to study enrolment
6. Medications or supplements that are known to alter gut function or microflora during the 4 weeks prior to study enrolment
7. Volunteers under anti-hyperlipidemic, antihypertensive, estrogen-related and/or anticoagulant agents
8. Prior gastrointestinal surgery (apart from appendectomy, cholecystectomy or herniotomy)
9. Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer.
10. Artificially sweetened beverage intake higher than 1000 ml/ per day
11. Female subjects will be excluded if they are pregnant, gave birth in the last 6 months, or are lactating.
12. Subject having a hierarchical or family link with the research team members.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Minimizing microbiota composition change | Daily from Day -4 to day + 7 (Day 0 is the start of the challenge)
  Shotgum metagenomics

SECONDARY OUTCOMES:
Increased intestinal microbiota diversity | Daily from Day -4 to day + 7 (Day 0 is the start of the dietary challenge)
  Measured by the Shannon diversity index
Increased microbiota gene richness | Daily from Day -4 to day + 7 (Day 0 is the start of the dietary challenge)
  Measured by gene counts from metagenome sequencing of the fecal microbiota
Gut comfort | Daily from Day -10 to day + 7 (Day 0 is the start of the dietary challenge)
  Assessed each Gastrointestinal Symptoms (VOMITING, NAUSEA, AUDIBLE BOWEL SOUNDS, FLATULENCE, ABDOMINAL CRAMPS, BLOATING ) with a scale (from 0 to 10, 10 being the worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Sami Damak, Principal Investigator — Société des produits Nestlé
Locations (1):
- Société des produits Nestlé/Metabolic Unit, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No